CLINICAL TRIAL: NCT03018743
Title: Discontinuation of Dapoxetine Treatment in Patients With Premature Ejaculation: a 2-year Prospective Observational Study
Brief Title: Discontinuation of Dapoxetine Treatment in Patients With Premature Ejaculation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jun Park, Associate Professor, Pusan National University Hospital
Other Study IDs: PNU-Dapoxetine
Record Dates: First submitted 2017-01-08; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — dapoxetine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dapoxetine treatment group: Consecutive patients who seek medical treatment for PE will be enrolled in the study.
  Interventions: Drug: Dapoxetine

INTERVENTIONS:
Drug: Dapoxetine — Patients receive dapoxetine (taken 1-3 hours before sexual intercourse) 30mg as needed. A dose escalation to 60mg will be consented after 1 month in case of low efficacy. Patients will be re-evaluated 1, 3, 6, 12, and 24 months after initiating therapy regarding the treatment status and the reasons for treatment discontinuation in the case of discontinuation. If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.
  Other Names: Priligy

SUMMARY:
Premature ejaculation (PE) has been known as one of the most common male sexual dysfunction.

Until now dapoxetine is the only approved medical treatment option and there is no second line therapy in case of no-response or refuse to dapoxetine, a comprehensive evaluation of the factors that lead to dropout is needed especially in a real-practice setting.

With this background, investigators are going to assesse the discontinuation rate of dapoxetine treatment in patients with PE and the reasons for discontinuation in a clinical setting throughout a follow-up period of 2 years.

DETAILED DESCRIPTION:
Premature ejaculation (PE) has been known as one of the most common male sexual dysfunction. PE can deteriorate sexual satisfaction and quality of life of the patients and their partners. Recently, the International Society for Sexual Medicine (ISSM) gave a definition that PE is a 'male sexual dysfunction characterized by ejaculation that always or nearly always occurs prior to or within 1 min of vaginal penetration from the first sexual experience (lifelong PE), or a clinically significant reduction in latency time, often to about 3 min or less (acquired PE)' . Until now, several treatment modalities for PE have been introduced. Psychological/behavioral; pharmacologic therapies, including selective serotonin reuptake inhibitors (SSRIs), tricyclic antidepressants, tramadol, phosphodiesterase 5 inhibitor, alpha 1-andreoreceptor antagonists; topical anaesthetics, and even surgical treatments have been used for PE in practice. Dapoxetine is the first oral pharmacological agent developed for the treatment of PE and the only SSRI approved in more than 60 countries for PE. The introduction of dapoxetine was accompanied with high expectation because of the optimal efficacy/ safety profile showed in the phase 3 trials. However, several clinical studies using depoxetine confirmed the efficacy in increasing IELT, it reveals significant dropout rate likely which was shown in the treatment using off-label SSRIs. Despite high efficacy and safety, discontinuation rate of dapoxetine is high compared to PDE5 inhibitors in patients with erectile dysfunction (ED).

Until now dapoxetine is the only approved medical treatment option and there is no second line therapy in case of no-response or refuse to dapoxetine, a comprehensive evaluation of the factors that lead to dropout is needed especially in a real-practice setting. With this background, investigators will assesse the discontinuation rate of dapoxetine treatment in patients with PE and the reasons for discontinuation in a clinical setting throughout a follow-up period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* men without history of dapoxetine treatment;
* > 19 years old; and involvement in a stable,
* monogamous relationship with a female sexual partner

Exclusion Criteria:

* penile anatomical deformity;
* spinal cord injury;
* radical prostatectomy;
* pelvic organ surgery;
* diagnosis of another sexual disorder except ED;
* an uncontrolled psychiatric disorder;
* history of major hematological, renal, or hepatic abnormalities;
* a history of alcoholism or substance abuse;
* organic illness causing limitations in assuming SSRIs

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients who seek medical treatment for PE will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Discontinuation rate of dapoxetine treatment | 1 month after initiating therapy
  Patients will be evaluated 1 month after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.
Discontinuation rate of dapoxetine treatment | 3 months after initiating therapy
  Patients will be evaluated 3 months after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.
Discontinuation rate of dapoxetine treatment | 6 months after initiating therapy
  Patients will be evaluated 6 months after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.
Discontinuation rate of dapoxetine treatment | 12 months after initiating therapy
  Patients will be evaluated 12 months after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.
Discontinuation rate of dapoxetine treatment | 24 months after initiating therapy
  Patients will be evaluated 24 months after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.

SECONDARY OUTCOMES:
Reasons of discontinuation of dapoxetine treatment | 1 month after initiating therapy
  Patients will be evaluated 1 month after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  The secondary outcome measures are the reasons of discontinuation of dapoxetine treatment (ex, high cost, low efficacy, side effects, etc)
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.
Reasons of discontinuation of dapoxetine treatment | 3 months after initiating therapy
  Patients will be evaluated 3 months after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  The secondary outcome measures are the reasons of discontinuation of dapoxetine treatment (ex, high cost, low efficacy, side effects, etc)
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.
Reasons of discontinuation of dapoxetine treatment | 6 months after initiating therapy
  Patients will be evaluated 6 months after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  The secondary outcome measures are the reasons of discontinuation of dapoxetine treatment (ex, high cost, low efficacy, side effects, etc)
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.
Reasons of discontinuation of dapoxetine treatment | 12 months after initiating therapy
  Patients will be evaluated 12 months after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  The secondary outcome measures are the reasons of discontinuation of dapoxetine treatment (ex, high cost, low efficacy, side effects, etc)
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.
Reasons of discontinuation of dapoxetine treatment | 24 months after initiating therapy
  Patients will be evaluated 24 months after initiating therapy regarding the treatment status (whether they treat or drop-out) for treatment discontinuation in the case of discontinuation.
  The secondary outcome measures are the reasons of discontinuation of dapoxetine treatment (ex, high cost, low efficacy, side effects, etc)
  If patients missed any visits, they will be contacted by telephone or mail to collect their treatment data.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No